CLINICAL TRIAL: NCT01464242
Title: Therapeutic Gain of Adding the Immunomodulator Pentoxifylline to the Treatment of Cutaneous Leishmaniasis
Brief Title: Add-on Study of Pentoxifylline in Cutaneous Leishmaniasis
Acronym: GT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centro Internacional de Entrenamiento e Investigaciones Médicas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 222951928964
Record Dates: First submitted 2011-10-24; First posted 2011-11-03 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Cutaneous Leishmaniasis; pentoxifylline; immunomodulation
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Meglumine Antimoniate; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucantime® + pentoxifylline (Experimental): Glucantime® 20mg/kg/day intramuscular injection (IM) daily for 20 days + pentoxifylline 400mg orally 3 times a day for 20 days.
  Interventions: Drug: Meglumine antimonate; Drug: Pentoxifylline
- Glucantime® + placebo (Placebo Comparator): Glucantime® 20mg/kg/day IM each day for 20 days + placebo 400mg orally 3 times a day for 20 days.
  Interventions: Drug: Meglumine antimonate; Drug: Placebo

INTERVENTIONS:
Drug: Meglumine antimonate — Glucantime® 20mg/kg/day IM daily for 20 days
  Other Names: Glucantime ®
Drug: Placebo — Placebo 400mg orally 3 times a day for 20 days
  Arms: Glucantime® + placebo
Drug: Pentoxifylline — Pentoxifylline 400mg orally 3 times a day for 20 days
  Arms: Glucantime® + pentoxifylline

SUMMARY:
The purpose of this study is to determine whether adding pentoxifylline to treatment of American cutaneous leishmaniasis with meglumine antimoniate increases the rate and speed of clinical response without diminishing safety, and to identify immune correlates of the healing response.

DETAILED DESCRIPTION:
Failure of first line therapies for cutaneous leishmaniasis is a public health issue. Since pathogenesis of dermal leishmaniasis is mediated by the immune and inflammatory responses, resolution of disease and control of infection are intimately linked to the host response. Several investigations have substantiated "proof of principal" for the therapeutic gain of co-adjuvant immunotherapy. This study will evaluate the efficacy and safety of using pentoxifylline (PTX) as a co-adjuvant in the treatment of cutaneous leishmaniasis with meglumine antimoniate in a randomized, double-blind, controlled trial. One arm will receive meglumine antimoniate and PTX and the other arm will receive meglumine antimoniate plus placebo. Efficacy will be assessed at the end of the treatment, and 5, 7, 13 and 26 weeks after initiation of treatment. Efficacy will be measured as the proportion of patients with definitive cure at 26 weeks after initiation of treatment, and time to healing. Safety will be assessed at the end of treatment with respect to the frequency and severity of adverse events.

Blood samples will be taken to evaluate the effects of PTX invitro and ex vivo on cells of the immune system. Proliferation and secretion of cytokines relevant to the immune and inflammatory responses by peripheral blood mononuclear cells will be measured before and after treatment. Likewise, macrophages will be differentiated from peripheral blood monocytes and infected with a strain of L. panamensis transfected with the luciferase (luc) gene. The investigators will measure the capacity of patient macrophages to kill parasites before and after treatment using a luminometric assay of viable parasite burden. Additionally, the investigators will measure the expression of inducible nitric oxide synthase, an enzyme that is necessary for nitric oxide production, one of the main leishmanicidal mechanisms used by macrophages. The investigators postulate that the use of the co-adjuvant with antimonials will increase the therapeutic response and that indicators predictive of a healing response can be identified by this prospective analysis of the immune response and therapeutic outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of cutaneous leishmaniasis (parasitologic confirmation or presumptive biopsy plus a positive Montenegro skin test).
* Age between 18 and 65 years.
* Lesions of a duration equal to or greater than one month
* More than one lesion or single lesion greater than 3 cm in diameter.
* Willingness to participate in the study after being informed through a consent process approved by the institutional ethical review committee

Exclusion Criteria:

* Pregnant or lactating women, and women who are planning to conceive during the study or that reject the use of birth control methods.
* Medical conditions that compromise the immune system (HIV infection, neoplasias, diabetes mellitus, autoimmune diseases, or use of corticosteroids, immunomodulators or antineoplastic drugs).
* Medical conditions that preclude the use of antimonials or pentoxifylline (cardiac, renal, hepatic or pancreatic disease or abnormalities).
* Alcohol abuse or use of recreational drugs that interfere with adherence to treatment
* Use of drugs with antileishmanial potential during the previous 13 weeks, including pentavalent antimonials, amphotericin B, miltefosine, and pentamidine
* Use of Theophylline , anticoagulants or antiarrhythmics.
* Diffuse or disseminated leishmaniasis.
* Mucosal involvement secondary to Leishmania infection.
* Incapacity to attend the study visits or any other condition that according to the investigator could interfere with adherence to study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-11; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Primary efficacy outcome: Definitive Cure | Participants will be followed up to 26 weeks
  Definitive cure, defined as complete re-epithelialization and absence of inflammatory signs in all cutaneous leishmaniasis lesions, and absence of new leishmaniasis lesions
Primary safety outcome: Adverse Events | Participants will be followed up to 26 weeks
  Clinical and laboratory adverse events will be qualified according to the Common Toxicity Criteria for Adverse Effects (CTCAE). All unexpected non serious adverse events will be notified and expected adverse events of moderate or higher category will be reported. All serious adverse events will be reported.

SECONDARY OUTCOMES:
In vitro lymphoproliferation | Participants will be followed for an average of 20 days
  Proliferation of peripheral blood mononuclear cells (PBMCs) after stimulation invitro with L. panamensis antigens will be measured by tritiated thymidine uptake
Cytokine secretion by PBMCs | Participants will be followed for an average of 20 days
  Secretion of a panel of cytokines relevant to the inflammatory and immune responses will be measured in supernatants from PBMCs cultured with L. panamensis antigens using Luminex technology
Macrophage leishmanicidal capacity | Participants will be followed for an average of 20 days
  Macrophages will be differentiated from peripheral blood monocytes and their leishmanicidal capacity will be measured by luminometry after infecton with luciferase-transfected promastigotes.
Macrophage inducible nitric oxide synthase (iNOS) expression | Participants will be followed for an average of 20 days
  Macrophage expression of iNOS after infection will be measured by quantitative real-time Polymerase Chain Reaction (RT-PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Nancy C Saravia, PhD, Principal Investigator — Centro Internacional de Entrenamiento e Investigación Médica
Locations (1):
- Corporación Centro Internacional de entrenamiento e Investigaciónes Médicas, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Derived] Castro MDM, Cossio A, Velasco C, Osorio L. Risk factors for therapeutic failure to meglumine antimoniate and miltefosine in adults and children with cutaneous leishmaniasis in Colombia: A cohort study. PLoS Negl Trop Dis. 2017 Apr 5;11(4):e0005515. doi: 10.1371/journal.pntd.0005515. eCollection 2017 Apr. PMID 28379954